CLINICAL TRIAL: NCT06435546
Title: Adherence to Oral Therapies in Advanced Breast and Prostate Cancers: a Pilot Study
Brief Title: Adherence to Oral Therapies in Advanced Breast and Prostate Cancers
Acronym: AdOTAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-A00396-41
Record Dates: First submitted 2023-11-27; First posted 2024-05-30 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adherence oral anticancer therapies questionnaire (Experimental): Blood samples
  Interventions: Diagnostic Test: Blood samples; Other: Adherence to anti-cancer therapies questionnaires

INTERVENTIONS:
Diagnostic Test: Blood samples — Ferritin, Transferrin Saturation (TSAT), Serum iron, Haemoglobin, Albumin
Other: Adherence to anti-cancer therapies questionnaires — GIRERD questionnaire, AdOT questionnaire, Use of social networks and alternatives and complementary medicines using patient questionnaire, EORTC QLQC30, HADS, MNA, MSPSS

SUMMARY:
AdOTAC is a pilot study, open, prospective, single-center, one-arm. The 200 patients will be included. Patient is included at Day 0. The included patient will have the opportunity to complete the self-questionnaires either at the ICL on Day 0, or at home up to 10 days after the date of inclusion in the study. Blood samples are collected the day of enrolment (Day 0) in order to measure the following biological markers: ferritin, serum iron, TSAT, albumin, and haemoglobin, except if performed as part of routine care in the previous 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18 years old.
* Patient with inoperable advanced breast cancer treated with oral endocrine therapy and/or targeted therapy and patient with inoperable advanced prostate cancer treated with oral hormonal therapy and/or targeted therapy.
* Oral anticancer medications started for at least 3 months.
* With a performance status ≤ 3.
* Patient has understood, signed and dated the consent form.
* Patient covered by the social security system.

Exclusion Criteria:

* Patient with early breast cancer or localized prostate cancer.
* Patient with life expectancy < 3 months.
* Patient in progression
* Undergoing intravenous or oral cytotoxic chemotherapy (capecitabine, cyclophosphamide, vinorelbine).
* Patient who has not yet started oral anticancer therapies or who has started for less than 3 months.
* Patient unable to read or speak French.
* Patient already included in another therapeutic trial with an experimental molecule.
* Persons deprived of their liberty or under guardianship (including curatorship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-12-14 (Estimated); Study Completion 2027-06-04 (Estimated)

PRIMARY OUTCOMES:
Assess medication adherence to oral treatments in patients with advanced breast or prostate cancer. | one day
  Medication adherence to oral anticancer treatments will be assessed using a score based on the GIRERD adherence assessment (targeting oral anticancer treatments).
  The score is a scale ranging from 0 to 6 (good compliance = 6; poor compliance = 4 to 5; non-adherence ≤ 3).

SECONDARY OUTCOMES:
Identify if the performance status by the ECOG-PS score is associated with reduced adherence to oral anticancer treatments | one day
  The performance status by the ECOG-PS score (0 to 4).
Identify if comorbitities is associated with reduced adherence to oral anticancer treatments | one day
  Comorbidities using the Charlson score (0 to 37).
Identify if polypharmacy by the use of five or more medications apart from the current oral anti-cancer medications is associated with reduced adherence to oral anticancer treatments | one day
  Polypharmacy by the use of five or more medications apart from the current oral anti-cancer medications (0 to >5).
Identify if treatment regimen by a level of complexity is associated with reduced adherence to oral anticancer treatments | one day
  The treatment regimen by a level of complexity (4 levels) given by an oncologist.
Identify if biological markers are associated with reduced adherence to oral anticancer treatments | one day
  Biological markers (ferritin, TSAT, serum iron, haemoglobin, albumin) by a blood test.
Identify if sarcopenia is associated with reduced adherence to oral anticancer treatments | one day
  Sarcopenia by the body mass/fat mass ratio using imaging (SMI: skeletal muscle mass index).
Identify if quality of life using the EORTC-QLQ-C30 questionnaire score is associated with reduced adherence to oral anticancer treatments | one day
  Quality of life using the EORTC-QLQ-C30 questionnaire score.
Identify if Social and emotional support by the MSPSS questionnaire is associated with reduced adherence to oral anticancer treatments | one day
  Social and emotional support by the MSPSS questionnaire (Multidimensional Scale of Perceived Social Support) (12-35: low perceived support; 36-60: medium perceived support; 61-84: hugh perceived support)
Identify if HADS scale is associated with reduced adherence to oral anticancer treatments | one day
  Anxiety and/or depression using the Hospital Anxiety and Depression Scale (HADS).
  (If the score in a column is greater than or equal to 11, it means person suffer from anxiety or depression)
Identify if MNA is associated with reduced adherence to oral anticancer treatments | one day
  Malnutrition using the MNA (Mini-Nutritional Assessment) questionnaire (24-30 points: normal nutritional status; 17-23.5 points: at risk of malnutrition; less than 17 points: malnourished)
Identify if Use of social networks and alternatives and complementary medicines using patient questionnaire is associated with reduced adherence to oral anticancer treatments | one day
  Use of social networks and alternatives and complementary medicines using patient questionnaire developed specifically for the study population.
Assess medication adherence to oral treatments in patients with advanced breast or prostate cancer. | one day
  Medication adherence to oral anticancer treatments will also be assessed using the score from the new AdOT questionnaire. The score is a scale ranging from 0 (no adherence) to 100 (perfect adherence).
Study the relationship between the two adherence questionnaires. | one day
  Subgroup analysis by cancer type (breast; prostate), use of alternatives and complementary medicines (yes; no) and use of social media and networks (yes; no).
Describe and compare medication adherence to oral treatments | one day
  The correlation between the scores on the GIRERD and AdOT will be analysed.
Describe and compare patient characteristics (socio-demographic, clinical and contextual), medication adherence to oral anticancer treatments according to cancer type, use of alternative and complementary medicines and use of social media and networks. | one day
  Subgroup analysis by cancer type (breast; prostate), use of alternative and complementary medicines (yes; no) and use of social media and networks (yes; no).

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Massard, MD, Principal Investigator — Institut de Cancérologie de Lorraine; Naoual Boujedaini, PhD, Study Chair — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No